CLINICAL TRIAL: NCT06542276
Title: Single Vectored Thermal Pulsation Treatment in Patients Using Topical Immunomodulators in the Management of Dry Eye Disease
Brief Title: Single Lipiflow Treatment to Reduce Pharmacologic Burden in DED
Acronym: Reduce
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dunes Eye Consultants (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Steve Ferguson, Lead Optometrist/ Director of Dry Eye Treatment Center, Dunes Eye Consultants
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DunesEye
Record Dates: First submitted 2024-07-21; First posted 2024-08-07 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: MGD-Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Intervention Model Description: This study, known as the REDUCE study, was a prospective, non-randomized, single-site, non- comparative study that evaluated the efficacy of a single vectored thermal pulsation (VTP) treatment in patients who were currently being treated with topical immunomodulator agents. This study was conducted in compliance with the Declaration of Helsinski and was reviewed and approved by the WCG institutional review board (IRB). The study is registered in clinictrials.gov. All participants provided written informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Lipiflow treatment results (Other): A single thermal vectored pulsation treatment of MGD with 3 month results review of treatment to evaluate objective and subjective response.
  Interventions: Device: Thermal Vectored Pulsation

INTERVENTIONS:
Device: Thermal Vectored Pulsation — The LipiFlow® (Johnson & Johnson Vision, USA) Thermal Pulsation System, also known as vectored thermal pulsation, is a treatment that applies localized heat and pressure to the meibomian glands lining the eyelids. The device consists of a console connected to single-use, sterile devices applied to each eye known as activators. The activator includes an eye warmer with a large lens that gently sits on the conjunctiva of each eye. The activator cups the upper and lower eyelid and applies regulated, outward heat to the surface of the palpebral conjunctiva with an air bladder that intermittently provides directional, controlled massage of the eyelids to promote expression of the liquified contents.
  Other Names: Lipiflow

SUMMARY:
Purpose: To evaluate the efficacy of vectored thermal pulsation treatment in subjects with a history of dry eye disease currently using a topical immunomodulator medication.

DETAILED DESCRIPTION:
Prospective, non-randomized, interventional study. Subjects with bilateral use of a topical immunomodulator drop and a history of dry eye disease were recruited to participate. All subjects underwent a vectored thermal pulsation treatment (LipiFlow). Patients were seen at baseline in a visit immediately prior to treatment and at months 1 and 3 following treatment. Data collected included tear osmolarity, tear break up time (TBUT), tear meniscus height (TMH), meibomian gland function and patient-reported symptoms using the ocular surface disease index (OSDI) questionnaire. Following the 3-month visit, patients were given the option to resume topical immunomodulator therapy.

ELIGIBILITY:
Inclusion Criteria:

* No prior history of meibomian gland treatment procedures LipiFlow, TearCare, or I-Lux
* lifitegrast or cyclosporine eye drops daily for a period of at least one year but not exceeding five years
* Meibograpy documneted retention of at least 50% of meibomian glands.

Exclusion Criteria:

* evidence of meibomian gland dropout exceeding 50%
* ocular rosacea,
* ocular surgery within the preceding three months
* prior in-office thermal meibomian gland treatment
* ocular trauma within preceding three months
* ocular herpetic infection
* chronic or recurrent inflammation
* eyelid abnormalities affecting lid function ocular surface abnormalities compromising corneal integrity (eg, epithelial basement membrane dystrophy, corneal burn)
* pregnant

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects discontinuing Topical Immunomodulator use | 3 months
  OSDI, TBUT, Tear Osmolarity, Meibomian gland expression quantity, TM

CONTACTS AND LOCATIONS:
Locations (1):
- Dunes Eye Consultants, Dakota Dunes, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Yes
Abstract
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 12months
Access Criteria: website
URL: https://www.duneseye.com